CLINICAL TRIAL: NCT03499834
Title: A Phase II Study to Evaluate the Safety and Efficacy of Ex Vivo Expanded Autologous Immune Killer Cells (IKC) in Stage IV Non-small Cell Lung Cancer (NSCLC) in Patients Who Failed Chemotherapy or Target Therapy
Brief Title: A Study to Evaluate the Safety and Efficacy of Ex Vivo Expanded Autologous Immune Killer Cells (IKC) in Stage IV Non-small Cell Lung Cancer (NSCLC) in Patients Who Failed Chemotherapy or Target Therapy
Acronym: IVY03
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ivy Life Sciences, Co., Ltd (Industry)
Collaborators: Taipei Veterans General Hospital, Taiwan (Other Government); Tri-Service General Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IVY03
Record Dates: First submitted 2018-04-02; First posted 2018-04-17 (Actual); Last update posted 2020-04-16 (Actual); Status verified 2020-04

CONDITIONS: Non-small Cell Lung Cancer (NSCLC) Stage IV
Keywords: Immune Cell Therapy; IKC
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Study Group (Experimental): 26 patients who has successfully undergone the screening criteria will be enrolled for treatment. Immune Killer Cells (IKC) will be administered through Intravenous Injection (I.V.) Frequency: One injection per week, twenty-four injections on-treatment
  Interventions: Biological: Immune Killer Cells (IKC)

INTERVENTIONS:
Biological: Immune Killer Cells (IKC) — Autologous cells of the immune system. Intravenous Injection (I.V.) frequency: One injection per week, twenty-four injections on-treatment

SUMMARY:
In this study, whole blood is drawn from the patient to be used to grow Immune Killer Cells (IKC). After proliferation, the IKC will be infused back into the patient to treat the cancer for a total of 24 weekly treatments.

Possible adverse reaction can include slight fever and headache.

ELIGIBILITY:
Inclusion Criteria:

1. Age≧20 years old
2. Life expectancy≧3 months
3. Eastern Cooperative Oncology group (ECOG) score 0~2
4. Cytologically-or histologically-confirmed non-small cell lung cancer（NSCLC)
5. Patients with clinical TNM classification of Malignant Tumours (TNM) stage IV...

Exclusion Criteria:

1. Patients with history of cardiovascular disease, including uncontrolled hypertension, congestive heart failure, myocardial infarction, angina pectoris, coronary artery disease, uncontrolled arrhythmia , previous history of encephalopathy within the past six months of screening period
2. Patients with HIV, HTLV or active tuberculosis
3. Women who are pregnant or breast-feeding
4. Patients with drug or other substance abuse
5. Patients with any other major disease, serious organ failure or patients unfit for participating in the trial (by the investigator's judgment)

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2017-12-05 (Actual); Primary Completion 2020-02-16 (Actual); Study Completion 2020-02-16 (Actual)

PRIMARY OUTCOMES:
Progression-Free Survival (PFS) | 6 months
  The length of time during and after the treatment of a disease, that a patient lives with the disease but it does not get worse

SECONDARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events [Safety] | 7 months
  Adverse Events (AE) and Serious Adverse Events (SAE) according to National Cancer Institute Criteria for Common Terminology Criteria for Adverse Events version 4.03 (NCI CTCAE v4.03) will be recorded and evaluated for their relationship to the treatment
Quality of Life (QOL) | 8 months
  The assessment will be performed using The World Heath Organization Quality of Life Questionnaire (WHOQOL)
  This questionnaire produces a quality of life profile. It is possible to derive four domain scores. The four domain scores denote an individual's perception of quality of life in each particular domain (1. Physical health 2. Psychological 3. Social relationships 4. Enviromental) Domain scores are scaled in a positive direction (i.e. higher scores denote higher quality of life).
  The mean score of items within each domain is used to calculate the domain score (min: 0 max: 100)
  Domain scores are then calculated (divide domain score by 4) to produce a final QOL Score (i.e. higher scores denote higher quality of life min: 0 max:100).

CONTACTS AND LOCATIONS:
Overall Officials: Yuh-Min Chen, MD, PhD, Principal Investigator — Taipei Veterans General Hospital, Taiwan
Locations (2):
- Taiwan (2):
  - Taipei Veterans General Hospital, Taipei
  - Tri Service General Hospital, Taipei

REFERENCES:
- [Derived] Tseng YH, Ho CL, Chian CF, Chiang CL, Chao HS, Tsai CL, Perng WC, Hsiao CF, Chuang MH, Ko KH, Cheng YC, Chen SJ, Wang CJ, Chen YM. Immune killer cells treatment for previously treated stage IV NSCLC patients. Sci Rep. 2024 Aug 21;14(1):19374. doi: 10.1038/s41598-024-69587-x. PMID 39169058